CLINICAL TRIAL: NCT04993976
Title: Effects of Resistance Training in Mild to Moderate Clinically Frail Patients Awaiting Coronary Artery Bypass Graft.
Brief Title: Prehabilitation and Coronary Artery Bypass Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rec/00980 Wajeeha Sahar
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Coronary Artery Bypass Graft
Keywords: CABG; Fraility; Prehabilitation
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): Strength training along with warm-up and cool down for 8 weeks
  Interventions: Other: Resistant training (Prehabilitation)
- Control group (Active Comparator): Supervised Standard care plan for 8 weeks
  Interventions: Other: Active Comparator: Control group

INTERVENTIONS:
Other: Resistant training (Prehabilitation) — Resistance training (10-15 repetitions: major muscle groups of upper and lower limbs [eg, shoulder overhead press, biceps curl, knee lift, and quadriceps extension in sitting and hamstrings curl exercises], one to three sets each) for 20-60 minutes five days a week.
  Arms: Prehabilitation group
Other: Active Comparator: Control group — Conventional physiotherapy group followed basic pre-operative respiratory physiotherapy including deep breathing exercises, instructions in coughing techniques, mobilization, and active exercises of the upper limbs and thorax. Walk 30 m in the hospital ward.
  Arms: Control group

SUMMARY:
To evaluate the effects of Prehabilitation Resistance training on frailty and functional capacity in mild to moderate clinically frail patients awaiting Coronary Artery Bypass Grafting) CABG. This study will contribute to describing the effect of resistance training in mild to moderate frails patients and were directed to be the part of cardiac rehabilitation and define the effects of cardiac prehabilitation and to check whether the effects of resistance training or routine training is similar for quality of recovery in mild to moderate frails patients which undergone CABG.

DETAILED DESCRIPTION:
In literature, Coronary Artery Bypass Graft (CABG) is a form of heart surgery that redirects blood around clogged arteries to increase blood flow and oxygen to the heart. During CABG surgery, the surgeon uses a portion of a healthy vessel (either an artery or vein) from the leg, chest, or arm to create a bypass around the clogged artery. During CABG surgery with cardiopulmonary bypass, a heart-lung machine artificially maintains circulation blood and oxygenation while the surgeon operates on the heart. It includes exercise, lifestyle changes, education, and emotional support. It can help improve patient's health and enable them to live a more active life after the patient has had a heart attack or heart surgery or if the patient has long-term heart problems such as heart failure.

The time spent waiting for cardiac surgery to be scheduled is a period of great uncertainty for a patient. There appears to be heightened anxiety regarding the inclusion of physical activity in this time period, mainly as a result of their current cardiac condition or diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective primary isolated coronary artery bypass grafting,

  * Patients with double and triple-vessel coronary artery disease.
  * Mild to moderately frail patients with a clinical frailty score of 5 -6 at the time of accepting surgery at the outpatient cardiothoracic surgical clinic.

Exclusion Criteria:

* Patient with musculoskeletal disability and neurological disability affecting respiratory rate.

  * Patient with renal dysfunction requiring dialysis, use of immunosuppressive treatments during the 30-day period before surgery,
  * Left ventricular ejection fraction <30%
  * concomitant valve disease
  * Patient having dysrhythmias or pacemaker dependent
  * Those patients who are severely frail (CFS 7-9)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Frailty | 8 weeks
  It is a scale ranges from 1 (very fit) to 9 (terminally ill). with common cut-off categories classified as non-frail (scores 1-3), vulnerable/ pre-frail (score 4) and frailty (scores 5-9). it is a simple, quick and highly predictive semi-quantitative tool.

SECONDARY OUTCOMES:
Functional capacity | 8 weeks
  It is measured through six minute walk test which is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Faisalabad Institute of Cardiology., Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afilalo J, Lauck S, Kim DH, Lefevre T, Piazza N, Lachapelle K, Martucci G, Lamy A, Labinaz M, Peterson MD, Arora RC, Noiseux N, Rassi A, Palacios IF, Genereux P, Lindman BR, Asgar AW, Kim CA, Trnkus A, Morais JA, Langlois Y, Rudski LG, Morin JF, Popma JJ, Webb JG, Perrault LP. Frailty in Older Adults Undergoing Aortic Valve Replacement: The FRAILTY-AVR Study. J Am Coll Cardiol. 2017 Aug 8;70(6):689-700. doi: 10.1016/j.jacc.2017.06.024. Epub 2017 Jul 7. PMID 28693934
- [Background] Sepehri A, Beggs T, Hassan A, Rigatto C, Shaw-Daigle C, Tangri N, Arora RC. The impact of frailty on outcomes after cardiac surgery: a systematic review. J Thorac Cardiovasc Surg. 2014 Dec;148(6):3110-7. doi: 10.1016/j.jtcvs.2014.07.087. Epub 2014 Aug 7. PMID 25199821
- [Background] Stammers AN, Kehler DS, Afilalo J, Avery LJ, Bagshaw SM, Grocott HP, Legare JF, Logsetty S, Metge C, Nguyen T, Rockwood K, Sareen J, Sawatzky JA, Tangri N, Giacomantonio N, Hassan A, Duhamel TA, Arora RC. Protocol for the PREHAB study-Pre-operative Rehabilitation for reduction of Hospitalization After coronary Bypass and valvular surgery: a randomised controlled trial. BMJ Open. 2015 Mar 9;5(3):e007250. doi: 10.1136/bmjopen-2014-007250. PMID 25753362
- [Background] Afilalo J, Kim S, O'Brien S, Brennan JM, Edwards FH, Mack MJ, McClurken JB, Cleveland JC Jr, Smith PK, Shahian DM, Alexander KP. Gait Speed and Operative Mortality in Older Adults Following Cardiac Surgery. JAMA Cardiol. 2016 Jun 1;1(3):314-21. doi: 10.1001/jamacardio.2016.0316. PMID 27438112
- [Derived] Sahar W, Waseem M, Riaz M, Nazeer N, Ahmad M, Haider Z. Effects of prehabilitation resistance training in mild to moderate clinically frail patients awaiting coronary artery bypass graft surgery. J Investig Med. 2024 Jan;72(1):151-158. doi: 10.1177/10815589231207795. Epub 2023 Oct 30. PMID 37804162